CLINICAL TRIAL: NCT01094444
Title: Placebo-controlled Trial Investigating the Effect of Vitamin K3-lotion for the Treatment of Cetuximab Induced Folliculitis
Brief Title: Investigation of the Effect of Vitamin K3-lotion for the Treatment of Cetuximab Induced Folliculitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Per Pfeiffer (Other)
Responsible Party: Sponsor-Investigator, Per Pfeiffer, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09.15
Record Dates: First submitted 2010-02-22; First posted 2010-03-29 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Folliculitis
Keywords: Vitamin K3 lotion; Cetuximab induced folliculitis
MeSH Terms: conditions — Folliculitis | interventions — Vitamin K 3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin K3-lotion (Experimental): A lotion containing 1.5 mM Vitamin K3.
  Interventions: Other: Vitamin K3
- B (No Intervention): Standard lotion without Vitamin K3

INTERVENTIONS:
Other: Vitamin K3 — Lotion containing 1.5 mM Vitamin K3
  Arms: Vitamin K3-lotion

SUMMARY:
The study aims to explore the benefit of topical vitamin K3 lotion for the reactivation/rephosphorylation of EGF-receptor in the skin and the possible reduction in cutaneous side effects of EGFr-inhibition.

Primary aim: The possible reduction of cutaneous side effects: folliculitis, dryness and redness of the skin.

Secondary aim: To explore any possible side effects of topical vitamin K3 lotion.

Methods: 36 patients with metastatic colorectal cancer or metastatic head and neck cancer allocated to treatment with chemotherapy and biweekly cetuximab. Two equally sized areas of at least 10x10 cm on the back or chest of the patient is marked. Patients receive in a double blinded procedure placebo lotion on one side and vitamin K3 lotion on the other side. The treatment may last for a maximum of two months and the patients are followed biweekly with photos, VAS-scores, questionnaires and CTCAE estimations. The patient will be able to take weekly photos at home during the weeks they are not seen at the outpatient clinic. During the treatment all other skin products or antibiotics is allowed and will be carefully registered by the health care professionals in the outpatient clinic.

The patient may enter the trial in two different ways: 18 patients start treatment with study lotions at the time they start treatment with cetuximab. The other 18 patients start treatment with study lotions when folliculitis appears.

Patients are asked for 1.5 mm skin biopsies of both study areas of the skin before start of treatment and after 4 weeks of treatment with placebo lotion and vitamin K3 lotion. These biopsies will be investigated for EGFr, phosphorylated EGFr and other central downstream mechanisms. The biopsy part of the study is optional for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Planned or ongoing treatment with cetuximab
* Age at least 18 years
* Informed written consent according to local and national legislation

Exclusion Criteria:

* Known disease that can influence either treatment, evaluation and the outcome of the current disease and treatment, including chronic dermatology
* Known hypersensitivity to menadion
* Concomitant treatment with Vitamin K or Vitamin K-antagonists
* Known psychological, family, sociological or geographic conditions which potentially can influence planned study treatment or follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Potential reduction in skin toxicity by vitamin K3 lotion | 3 months
  Reduction in numbers of papulo-pustular eruptions in the treatment fields. Changes in follicular eruptions, dryness/redness of skin estimated by CTCAE 4.0. Patients own experience of efficacy estimated by questionaire and VAS scale.

SECONDARY OUTCOMES:
Potential toxicity of vitamin K3 lotion | 3 months
  No systemic or skin toxicity is expected. Therefore all experienced skin changes will be estimated by CTCAE 4.0. Furthermore, broad bloodtest screenings will be done bi-weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper G. Eriksen, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

REFERENCES:
- [Background] Eriksen JG, Kaalund I, Clemmensen O, Overgaard J, Pfeiffer P. Placebo-controlled phase II study of vitamin K3 cream for the treatment of cetuximab-induced rash. Support Care Cancer. 2017 Jul;25(7):2179-2185. doi: 10.1007/s00520-017-3623-x. Epub 2017 Feb 15. PMID 28197850